CLINICAL TRIAL: NCT05201729
Title: Exploring the Influence Factors of the Efficacy of PD-1 Monoclonal Antibody Therapy in Advanced Pancreatic Cancer After Failure of First-line Chemotherapy by Using Multiomics Technology
Brief Title: Influence Factors of PD-1 Therapeutic Efficacy in Advanced Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, duowu zou, Chief physician, Ruijin Hospital
Other Study IDs: RJ2020368
Record Dates: First submitted 2022-01-10; First posted 2022-01-21 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma, PDAC
MeSH Terms: conditions — Anophthalmia with pulmonary hypoplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — n situ tissue samples of pancreatic cancer by EUS-FNAare immediately sent to the laboratory for sequencing.
  Serum, plasma and peripheral blood mononuclear cells (PBMC) are isolated from peripheral blood samples; Serum and plasma are stored in - 80 ℃ refrigerator, and PBMC are stored in liquid nitrogen.
  Biological samples of all patients are kept in a regulated biological sample bank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The early diagnosis rate of pancreatic cancer is low and most patients rely on palliative chemotherapy. However, the clinical benefit and objective response rate (ORR) of patients with first-line chemotherapy are low. Therefore,it is essential to develop new therapies to improve the survival of patients with pancreatic cancer.

DETAILED DESCRIPTION:
In this study, patients with advanced pancreatic cancer who failed in the first-line chemotherapy will be included to receive anti-PD-1 monoclonal antibody treatment, and a high-throughput study with a small sample size will be carried out by using multiomics technology to capture the heterogeneity of response to PD-1 therapy in patients with pancreatic cancer.The investigators choose two time points: after chemotherapy failure (before PD-1 therapy) and during efficacy evaluation（after PD-1 therapy）, to obtain in situ samples of pancreatic cancer tissues by EUS-FNA.The samples are tested by dynamic multi-omics studybefore and after treatment (including genomics, transcriptomics, metabonomics, proteomics, etc.).And combining the results with the drug reaction and clinical outcome of patients for a comprehensive analysis.The purpose of this study is to explore the potential biomarkers or omics of PD-1 therapy and lay the foundation for building a model to predict the effect of PD-1 therapy in patients with advanced pancreatic cancer.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

1. Age > 18 years old, male or female;
2. Locally advanced or metastatic pancreatic ductal adenocarcinoma confirmed by histopathology / cytology of the primary and / or metastatic lesions and unsuitable for surgical resection;
3. The failure of first-line chemotherapy with gemcitabine or FOLFINOX, disease progression or intolerable severe toxicity;
4. The time from the end of the last chemotherapy should be more than 28 days;
5. According to the evaluation criteria of solid tumor efficacy(RECIST 1.1), there should be at least one measurable lesion (non nodular lesion with the longest diameter of 210 mm, or nodular lesion with the shortest diameter of more than 15 mm);
6. ECOG score:0~2;
7. Hematology, biochemistry and organ function indexes meet the following requirements:

   * The absolute count of neutrophils (ANC) is more than 1.5x10% / L
   * Platelet count (PLT) ≥ 80x109/l
   * Hemoglobin (HB) ≥ 9.0 g/dl
   * TBIL is less than 2.0 ULN, albumin (ALB) 230g / L
   * In patients without liver metastasis, alanine transaminase (ALT) and / or aspartate -transaminase (AST) are less than 3.0 ULN
   * Patients with liver metastasis, ALT and / or ASTS <5.0*ULN
   * Serum creatinine (CREA) < 1.5 x ULN, and creatinine clearance rate (CER) ≥ 30ml / min (Cockcroft-Gault);
8. Women of childbearing age receives negative pregnancy test within 14 days before treatment. Male and female patients of childbearing age and their sexual partners agree to use reliable contraceptive methods within 14 days before enrollment, during the study and within 60 days after drug withdrawal；
9. Patients voluntarily participate in this study, sign informed consent, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

If any of the following criteria is met, the patient should be excluded:

1. Pancreatic ductal adenocarcinoma is diagnosed without histopathology / cytology;
2. The target lesion has received local non-drug therapy (including radiotherapy, physical and / or chemical ablation, etc.), and there is no imaging progression;
3. If the central nervous system metastasis is known, MRI should be performed to exclude it;
4. Patients with carcinoma of Vater's ampulla or adenocarcinoma of biliary tract;
5. Patients with partial or complete intestinal obstruction or complete biliary obstruction that cannot be relieved by active treatment;
6. Ascites increases gradually after 2 weeks of conservative treatment (such as diuresis, sodium restriction, excluding ascites drainage);
7. In the past 5 years, patients had a history of other malignant tumors, except for the following two cases: a)After other malignant tumors treated by a single operation, 5-year disease-free survival (DFS) was achieved;b)Cured basal cell carcinoma of the skin and cured carcinoma in situ of the cervix;
8. Pregnant or lactating women;
9. Active infection; Poorly controlled hypertension (≥ 150 / 100mmhg); Angina pectoris and unstable angina pectoris in recent 3 months, myocardial infarction, cardiac insufficiency (> NYHA class II), schizophrenia, or history of psychotropic drug abuse in 1 year before enrollment;
10. If HBV-DNA is more than 104 copies or more than 2000 IU / ml, antiviral and liver protection therapy should be carried out first. Only when HBV-DNA is less than 104 copies (2000 IU / ml), can the patients be enrolled in the group, and continue to take antiviral drugs, monitor liver function and HBV viral load; HCV antibody or HCV-RNA were positive; HIV infected patients (non high risk group, without clinical symptoms or signs indicating HIV infection, HIV test may not be carried out);
11. Any of the following treatments were given within prior to enrollment:

    1. Within 4 weeks, received surgery of grade II or above (according to the operation classification catalogue (revised version in 2014) issued by the state health and Family Planning Commission); No matter whether it is related to tumor or not);
    2. Received extended radiotherapy within 4 weeks or limited range radiotherapy within 2 weeks (researchers in each center can judge the appropriate time to enter the group according to the recovery of toxicity after radiotherapy);
    3. Within 4 weeks or participating in other therapeutic / interventional clinical trials;
    4. Received local anti-tumor therapy within 4 weeks;
12. NCI ctcae2 or above toxicity caused by previous treatment and not yet recovered (excluding hair loss and skin pigmentation);
13. It is known that PD-1 monoclonal antibody and its excipients are allergic or intolerable;
14. There are other situations that the researchers think are not suitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced pancreatic cancer who failed in the first-line chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference of progression free survival (PFS) | 1.5 years
  The time from random to the first occurrence of disease progression or death from any cause.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 1.5 years
  The percentage of cases with remission and disease stability after treatment in the whole evaluable cases.
the quality of participants'life | 1.5 years
  According to the European Organization for research and treatment of cancer (EORTC) quality of life core scale EORTC QLQ-C30 (V3.0 Chinese version)，evaluating the quality of life (QOL)

CONTACTS AND LOCATIONS:
Overall Officials: Duowu Zou, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China